CLINICAL TRIAL: NCT05301309
Title: The Effects of Integrative Early Breastfeeding Support and Intervention Program on Preterm Infants' Breastfeeding Rate and Neurobehavioral Development and Maternal Mental Health
Brief Title: Integrative Early Breastfeeding Support in NICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 202106048RIND
Record Dates: First submitted 2022-02-28; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-02

CONDITIONS: Premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding Consultation (Experimental): The intervention group would receive integrative early breastfeeding support and intervention programs, including "breastfeeding for prematurity brochure", group education class, weekly interview, one-by-one breastfeeding consultation and online peer group support.
  Interventions: Behavioral: breastfeeding consultation
- routine care (Active Comparator): The control group only receive "breastfeeding for prematurity brochure" and routine care.
  Interventions: Behavioral: breastfeeding consultation

INTERVENTIONS:
Behavioral: breastfeeding consultation — Integrative early breastfeeding support and intervention programs: breastfeeding for prematurity brochure, group education class, weekly interview, one-by-one breastfeeding consultation and online peer group support.

SUMMARY:
Background and Purpose: Preterm infants are suffered from preterm-related medical sequelae and neurobehavioral problems, which required interdisciplinary intervention. Breast milk is the best nutrition for preterm infants. However, consistent breastfeeding is quite challenging to most mothers of prematurity. The purpose of this study is to investigate the effect of integrative early breastfeeding support and intervention programs on preterm infants' breastfeeding rate, neurobehavioral development, and maternal mental health. Method: The prospective, single-blinded randomized controlled trial would be conducted in National Taiwan University Children's Hospital in Taipei, Taiwan. We would recruit the mother and infant dyad whose gestational age is between 28 weeks and 34 6/7 weeks. The intervention group (n=22) would receive integrative early breastfeeding support and intervention programs, including breastfeeding for prematurity brochure, group education class, weekly interview, one-by-one breastfeeding consultation and online peer group support. The control group (n=22) only receive breastfeeding for prematurity brochure and routine care. Outcome measure: the growth date and types of feeding data at birth, discharge from hospital, 3- and 6-month-old of corrected age would be collected by medical chart review or by interview. Maternal health condition would evaluate by 3 questionnaires, including Breastfeeding Self-Efficacy Scale, Beck Depression Inventory-II and Maternal Confidence Questionnaire. Neurobehavioral development would be measured using Neonatal Neurobehavioral Evaluation-Chinese version and Bayley Scales of infant and toddler development 3rd edition at corrected age of 3-month-old and 6-month-old separately. Demographic data, birth history, types of breastfeeding data would be compared with independent t test or χ2 test. The effect of integrative early breastfeeding support and intervention on growth of preterm infants, neurobehavioral development, types of feeding, and maternal health would be conducted by logistic regression analysis.

DETAILED DESCRIPTION:
Preterm infants are suffered from preterm-related medical sequelae and neurobehavioral problems, which required interdisciplinary intervention. Breast milk is the best nutrition for preterm infants. However, consistent breastfeeding is quite challenging to most mothers of prematurity. The purpose of this study is to investigate the effect of integrative early breastfeeding support and intervention programs on preterm infants' breastfeeding rate, neurobehavioral development, and maternal mental health. Method: The prospective, single-blinded randomized controlled trial would be conducted in National Taiwan University Children's Hospital in Taipei, Taiwan. We would recruit the mother and infant dyad whose gestational age is between 28 weeks and 34 6/7 weeks. The intervention group (n=22) would receive integrative early breastfeeding support and intervention programs, including breastfeeding for premature brochure, group education class, weekly interview, one-by-one breastfeeding consultation (at least once during admission) and online peer group support. The control group (n=22) only receive breastfeeding for premature brochure and routine care. Outcome measure: the growth data (including height, weight and head circumference) and types of feeding data at birth, discharge from hospital, 3- and 6-month-old of corrected age would be collected by medical chart review or by interview. Maternal health condition would evaluate by 3 questionnaires, including Breastfeeding Self-Efficacy Scale, Beck Depression Inventory-II and Maternal Confidence Questionnaire. Neuro-behavioral development would be measured using Neonatal Neurobehavioral Evaluation-Chinese version and Bayley Scales of infant and toddler development 3rd edition at corrected age of 3-month-old and 6-month-old separately. Demographic data, birth history, types of breastfeeding data would be compared with independent t test or χ2 test. The effect of integrative early breastfeeding support and intervention on growth of preterm infants, neurobehavioral development, types of feeding, and maternal health would be conducted by logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* the mother of preterm baby whose gestational age is between 28 weeks and 34 6/7 weeks.

Exclusion Criteria:

* mother less than 20-years-old
* not intend to breastfeed
* baby's vital sign is not stable the need frequent medical intervention
* baby had congenital anomaly, gene anomaly, neurological disease, mitochondrial disease or metabolic diseases
* mother or baby receive major surgery

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurobehavioral development | corrected age 3-month-old
  Neurobehavioral development was evaluated by Bayley-III
Neurobehavioral development | corrected age 6-month-old
  Neurobehavioral development was evaluated by Bayley-III

SECONDARY OUTCOMES:
body height | corrected age of 3-month-old
  baby's body height in centimetres
body height | corrected age of 6-month-old
  baby's body height in centimetres
body weight | corrected age of 3-month-old
  baby's body weight in grams
body weight | corrected age of 6-month-old
  baby's body weight in grams
head circumference | corrected age of 3-month-old
  baby's head circumference in centimetres
head circumference | corrected age of 6-month-old
  baby's head circumference in centimetres
Breastfeeding Self-Efficacy Scale | at birth
  Score of "Breastfeeding Self-Efficacy Scale", which minimum score is 14 and maximum score is 70. Higher scores mean better outcome.
Breastfeeding Self-Efficacy Scale | corrected age of 3-month-old
  Score of "Breastfeeding Self-Efficacy Scale", which minimum score is 14 and maximum score is 70. Higher scores mean better outcome.
Breastfeeding Self-Efficacy Scale | corrected age of 6-month-old
  Score of "Breastfeeding Self-Efficacy Scale", which minimum score is 14 and maximum score is 70. Higher scores mean better outcome.
Beck Depression Inventory-II | at birth
  Total score of "Beck Depression Inventory-II". The highest possible total for the test would be 63, and the lowest total of the test would be 0. Higher scores mean worse outcome.
Beck Depression Inventory-II | corrected age of 3-month-old
  Total score of "Beck Depression Inventory-II". The highest possible total for the test would be 63, and the lowest total of the test would be 0. Higher scores mean worse outcome.
Beck Depression Inventory-II | corrected age of 6-month-old
  Total score of "Beck Depression Inventory-II". The highest possible total for the test would be 63, and the lowest total of the test would be 0. Higher scores mean worse outcome.
Maternal Confidence Questionnaire | at birth
  Total score of "Maternal Confidence Questionnaire". The highest possible total for the test would be 70, and the lowest total of the test would be 14. Higher scores mean better outcome.
Maternal Confidence Questionnaire | corrected age of 3-month-old
  Total score of "Maternal Confidence Questionnaire". The highest possible total for the test would be 70, and the lowest total of the test would be 14. Higher scores mean better outcome.
Maternal Confidence Questionnaire | corrected age of 6-month-old
  Total score of "Maternal Confidence Questionnaire". The highest possible total for the test would be 70, and the lowest total of the test would be 14. Higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yu Yang, MSc, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No